CLINICAL TRIAL: NCT02930915
Title: Feasibility Study: Acquisition of Three Dimensional Facial Geometry of Patients' Scheduled for Head and Neck Radiotherapy Treatment.
Brief Title: Acquisition of 3D Facial Geometry of Patients' Scheduled for Radiotherapy Treatment
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of East Anglia (Other)
Collaborators: Clinical Research and Trials Unit (Norfolk & Norwich University Hospital, UK) (Other)
Responsible Party: Sponsor
Other Study IDs: 82-03-16
Record Dates: First submitted 2016-10-10; First posted 2016-10-12 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; Radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Hand-held laser scanner — The laser scanning is non-intrusive and the scan can be completed in approximately 15 minutes. The scanning process involves the patient sitting in a chair while a researcher performs the scan. As a precautionary measure we require the patient to wear an eye mask as although the scanner is CE marked and completely safe . The process can be completed in stages (e.g. 3 x 5 minutes) with a break of 2-3 minutes between each session. The laser scanner will then be moved around the patient to obtain a set of 3D points forming the surface of the patient's head. We believe the laser scanning to be the most accurate way to acquire the surface of the patient's face / head and we wish to compare the models we obtain with surfaces rendered from the patient's CT data set.

SUMMARY:
This study investigates the feasibility of using 3D-Printing to manufacture masks used to immobilize patients undergoing radiotherapy treatment for tumors affecting the head and neck.

DETAILED DESCRIPTION:
The current types of masks that are used in radiotherapy treatment sessions for those patients who have head-and-neck cancer are 'made to measure' and the methods currently employed to make them are invasive and in some cases patients' have found this to be particularly unpleasant. Their experience motivates research into less invasive and potentially more accurate techniques for their manufacture.

To effectively develop an automatic manufacturing pipeline, and to assess the accuracy of the approach we need access to CT data from a cohort of patients for which we also have an accurate (ground truth) 3D facial model. Such a model can be acquired in a few minutes using a hand-held laser scanner.

ELIGIBILITY:
Inclusion Criteria:

* Have a Head-and-neck cancer
* Receiving radiotherapy treatments (CT images)

Exclusion Criteria:

* Children (age less than 18)

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A cohort of patients who have a Head-and-neck cancer and receiving radiotherapy treatments in the Norfolk and Norwich University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
3D facial geometry of patient's head | 15 minutes
  The resultant 3D facial geometry of patient's head will be used to construct a 3D digital model which will be used to evaluate the accuracy of the model generated by CT images. In other words, the outcome will be used as a ground-truth for the CT-derived model.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Fisher, PhD, Principal Investigator — University of East Anglia
Locations (2):
- United Kingdom (2):
  - School of Computing Sciences, University of East Anglia, Norwich, Norfolk
  - Norfolk and Norwich Univeristy Hospital NHS foundation Trust, Norwich, Norfolk

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fisher, Mark, Christopher Applegate, Mohammad Ryalat, Stephen Laycock, Mark Hulse, Daniel Emmens, and Duncan Bell. Evaluation of 3-d printed immobilisation shells for head and neck IMRT. Open Journal of Radiology 4, no. 04 (2014): 322.
- [Background] Laycock, S. D., M. Hulse, C. D. Scrase, M. D. Tam, S. Isherwood, D. B. Mortimore, D. Emmens, J. Patman, S. C. Short, and G. D. Bell. Towards the production of radiotherapy treatment shells on 3D printers using data derived from DICOM CT and MRI: preclinical feasibility studies. Journal of Radiotherapy in Practice 14, no. 01 (2015): 92-98.